CLINICAL TRIAL: NCT05384093
Title: Outcomes of Treatment Using the ERMI Shoulder Flexionater®
Brief Title: Outcomes of Treatment Using the ERMI Shoulder Flexionater ®
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Collaborators: ERMI, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FORE AC 2019
Record Dates: First submitted 2022-05-03; First posted 2022-05-20 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Adhesive Capsulitis of Shoulder
MeSH Terms: conditions — Bursitis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Adhesive Capsulitis Study (Active Comparator): The purpose of this study is to compare treatment efficacy of patients with symptoms of primary and secondary adhesive capsulitis between three groups: 1) Patients treated with Physical Therapy alone; 2) Patients treated with the ERMI Shoulder Flexionater® alone; 3) Patients treated with PT + Device in the treatment.
  Interventions: Device: High Intensity Stretch Device
- Post operative Shoulder Stiffness Study (Active Comparator): The purpose of this study is to compare treatment efficacy of patients with post-operative stiffness indicative of secondary adhesive capsulitis between three groups: I) Patients treated with Physical Therapy alone; II) Patients treated with the ERMI Shoulder Flexionater® alone; III) Patients treated with PT + Device in the treatment.
  Interventions: Device: High Intensity Stretch Device
- Secondary Surgery Study (Active Comparator): The purpose of this study is to compare recovery of patients who have undergone a manipulation under anesthesia or a lysis of adhesions between three groups: 1) Patients treated with Physical Therapy alone; 2) Patients treated with the ERMI Shoulder Flexionater® alone; 3) Patients treated with PT + Device in the treatment.
  Interventions: Device: High Intensity Stretch Device

INTERVENTIONS:
Device: High Intensity Stretch Device — High Intensity Stretch and Physical Therapy are used either together or alone to treat study arm.
  Other Names: Physical Therapy

SUMMARY:
Study 1 - Adhesive Capsulitis Study - 110 patients The purpose of this study is to compare treatment of patients with symptoms of adhesive capsulitis, primary and secondary, between three groups: I) Physical Therapy alone; II) ERMI Shoulder Flexionater® alone; III) PT + Device.

Study 2 - Postoperative Shoulder Stiffness Study - 90 patients The purpose of this study is to compare treatment of patients with post-operative stiffness indicative of secondary adhesive capsulitis between three groups: I) Physical Therapy alone; II) ERMI Shoulder Flexionater® alone; III) PT + Device.

Study 3 - Stiffness after MUA Study - enroll all eligible patients (goal of at least 15) The purpose of this study is to compare treatment of patients who have undergone manipulation under anesthesia or lysis of adhesions between three groups: I) Physical Therapy alone; II) ERMI Shoulder Flexionater® alone; III) PT + Device.

DETAILED DESCRIPTION:
Study 1 - Adhesive Capsulitis Study (AC)

Objective: The purpose of this study is to compare treatment efficacy of patients with symptoms of primary and secondary adhesive capsulitis between three groups: 1) Patients treated with Physical Therapy alone; 2) Patients treated with the ERMI Shoulder Flexionater® alone; 3) Patients treated with PT + Device in the treatment.

1. Prospective randomized control trial
2. Sample size - 110 patients
3. Study Groups:

   1. Group I - Physical Therapy Only
   2. Group II - Flexionater® only
   3. Group III - Flexionater® and Physical Therapy
4. Length of study - 2-year follow-up from last enrolled patient

Study 2 - Postoperative Shoulder Stiffness Study (POS)

Objective: The purpose of this study is to compare treatment efficacy of patients with post-operative stiffness indicative of secondary adhesive capsulitis between three groups: I) Patients treated with Physical Therapy alone; II) Patients treated with the ERMI Shoulder Flexionater® alone; III) Patients treated with PT + Device in the treatment.

1. Prospective randomized control trial
2. Sample size - 90 enrolled patients
3. Study Groups:

   1. Group I - Physical Therapy only
   2. Group II - Flexionater® only
   3. Group III - Flexionater® and Physical Therapy
4. Length of study - 2-year follow-up from last enrolled patient

Study 3 - Secondary Surgery Study (SAM)

Objective: The purpose of this study is to compare recovery of patients who have undergone a manipulation under anesthesia or a lysis of adhesions between three groups: 1) Patients treated with Physical Therapy alone; 2) Patients treated with the ERMI Shoulder Flexionater® alone; 3) Patients treated with PT + Device in the treatment.

1. Prospective randomized control trial
2. Sample size - 10 enrolled patients
3. Study Groups:

   1. Group I Physical Therapy Only
   2. Group II - - Flexionater® only
   3. Group III - Flexionater® and Physical Therapy
4. Length of study - 2-year follow-up from last enrolled patient

ELIGIBILITY:
For Study Group 1- Adhesive Capsulitis (AC)

Inclusion Criteria:

* Exhibits symptoms of adhesive capsulitis i. Shoulder pain with limited motion for more than one month ii. AND ≤ 30 degrees external rotation with arm at side iii. AND ≤ 130 degrees forward flexion d. Cortisone shot for all patients

Exclusion Criteria:

* a. No prior shoulder surgery b. Infection c. Rheumatoid arthritis d. Any structural or systemic disorder that could result in pain or ROM limitation i. Such as inflammatory joint disease, osteoarthritis evidenced on radiographs ii. full thickness rotator cuff tear as shown by ultrasound imaging iii. history of major trauma or surgery involving the shoulder

For Study Group 2 - Postoperative Shoulder Stiffness Study (POS)

Inclusion Criteria:

c. Is not recovering normally based on objective criteria set for screening process i. Step 1 - Follow patients -all post-op patients with indicated procedures (see # 7 for list.) ii. Step 2 - Screen Patients -does patient meets inclusion criteria at 6 weeks or 3 months of follow-up?

1. < 15 degrees external rotation with arm at side at 6 weeks post-op
2. OR < 90 degrees forward flexion at 3 months post-op iii. Step 3 - Enroll patients that meet inclusion criteria and assign group

Exclusion Criteria:

a. Revision surgery b. Infection c. Rheumatoid arthritis

7. Procedures included

1. Shoulder arthroscopic procedures (29827, 29828, 29823,29824, 29826)
2. ORIF Humerus fracture (23615)

   For Study Group 3, Secondary Surgery Study (SAM)

   Inclusion Criteria:
3. Underwent a manipulation under anesthesia or a lysis of adhesions procedure

Exclusion Criteria:

a. Infection b. Rheumatoid arthritis c. Any structural or systemic disorder that could result in pain or ROM limitation i. Such as inflammatory joint disease, osteoarthritis evidenced on radiographs ii. full thickness rotator cuff tear as shown by ultrasound imaging iii. history of major trauma or surgery involving the shoulder

7. Procedures included

1. Manipulation under anesthesia (23700)
2. Lysis of adhesions (29825)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Shoulder Range of Motion Improvement | 3 months
  Measuring Shoulder External Rotation and Forward Flexion using a goniometer according to standard practice
Shoulder Range of Motion | 6 months
  Measuring Shoulder External Rotation and Forward Flexion using a goniometer according to standard practice
Shoulder Range of Motion | 12 months
  Measuring Shoulder External Rotation and Forward Flexion using a goniometer according to standard practice
Shoulder Range of Motion | 24 months
  Measuring Shoulder External Rotation and Forward Flexion using a goniometer according to standard practice
Shoulder Range of Motion | 6 weeks
  Measuring Shoulder External Rotation and Forward Flexion using a goniometer according to standard practice
Shoulder Range of Motion | baseline
  Measuring Shoulder External Rotation and Forward Flexion using a goniometer according to standard practice
VAS (Visual Analog Scale) Pain Score | 3 months
  Visual Analog Scale Pain Score 0 (no pain) - 10 (pain as bad as it can be)
VAS Pain Score | 6 weeks
  Visual Analog Scale Pain Score: 0 (no pain) - 10 (pain as bad as it can be)
VAS Pain Score | 6 months
  Visual Analog Scale Pain Score: 0 (no pain) - 10 (pain as bad as it can be)
VAS Pain Score | 12 months
  Visual Analog Scale Pain Score: 0 (no pain) - 10 (pain as bad as it can be)
VAS Pain Score | 24 months
  Visual Analog Scale Pain Score: 0 (no pain) - 10 (pain as bad as it can be)
VAS Pain Score | baseline
  Visual Analog Scale Pain Score: 0 (no pain) - 10 (pain as bad as it can be)
ASES Score | baseline
  American Shoulder and Elbow Society Score (10 activities of daily living are calculated)
ASES Score | 3 month
  American Shoulder and Elbow Society Score (10 activities of daily living are calculated)
ASES Score | 6 weeks
  American Shoulder and Elbow Society Score (10 activities of daily living are calculated)
ASES Score | 6 months
  American Shoulder and Elbow Society Score (10 activities of daily living are calculated)
ASES Score | 12 months
  American Shoulder and Elbow Society Score (10 activities of daily living are calculated)
ASES Score | 24 months
  American Shoulder and Elbow Society Score (10 activities of daily living are calculated)

SECONDARY OUTCOMES:
SST | Baseline
  Simple Shoulder Test
SST | 3 month
  Simple Shoulder Test
SST | 6 weeks
  Simple Shoulder Test
SST | 6 months
  Simple Shoulder Test
SST | 12 months
  Simple Shoulder Test
SST | 24 months
  Simple Shoulder Test
Device Compliance Questionnaire (if applicable) | 6 weeks
  compliance with Device usage
Device Compliance Questionnaire (if applicable) | 3 months
  compliance with Device usage
Device Compliance Questionnaire (if applicable) | 6 months
  compliance with Device usage

CONTACTS AND LOCATIONS:
Overall Officials: Peter Simon, PhD, Study Director — Foundation for Orthopaedic Research and Education
Locations (1):
- Foundation for Orthopaedic Research and Education, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
unknown at this time

REFERENCES:
- [Derived] Teytelbaum DE, Kumar NS, Dent CS, Neaville S, Warren DH, Simon P, Baker CE. Efficacy of a high-intensity home stretching device and traditional physical therapy in non-operative management of adhesive capsulitis - a prospective, randomized control trial. BMC Musculoskelet Disord. 2024 Apr 20;25(1):305. doi: 10.1186/s12891-024-07448-4. PMID 38643086